CLINICAL TRIAL: NCT03374280
Title: The Phase Three Trials of Pemetrexed/Cisplatin Intercalating Gefitinib vs Pemetrexed/Cisplatin Treating EGFR Wild NSCLC(Non Squamous Cell Carcinoma)
Brief Title: Pemetrexed/Cisplatin Intercalating Gefitinib Treating EGFR Wild NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Haihong Yang, MD, Pricipal investigator, Chief Physician, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangzhouMC
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; Gefitinib; EGFR negative; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pemetrexed/cisplatin intercalating gefitinib (Experimental): pemetrexed 500mg/m2 d1; cisplatin 30mg/m2 d1-2 ;gefitinib 250mg d3-20d, to 4 cycles.
  pemetrexed 500mg/m2 d1; gefitinib 250mg d2-20d to disease progression or untolerable
  Interventions: Drug: pemetrexed/cisplatin intercalating gefitinib
- pemetrexed/cisplatin (Active Comparator): pemetrexed 500mg/m2 d1; cisplatin 30mg/m2 d1-2 to 4 cycles. pemetrexed 500mg/m2 d1 to disease progression or untolerable
  Interventions: Drug: pemetrexed/cisplatin

INTERVENTIONS:
Drug: pemetrexed/cisplatin intercalating gefitinib
  Arms: pemetrexed/cisplatin intercalating gefitinib
Drug: pemetrexed/cisplatin
  Arms: pemetrexed/cisplatin

SUMMARY:
To investigate the curative effect between Pemetrexed/Cisplatin and Pemetrexed/Cisplatin intercalating Gefitinib Treating EGFR Wild NSCLC

DETAILED DESCRIPTION:
In preclinical data, it is identified that pemetrexed combined with erlotinib could achieve good response than pemetrexed because EGFR-TKI (erlotinib) could enhance the sensitivity of pemetrexed. So we design the trial to investigate curative effect between Pemetrexed/Cisplatin and Pemetrexed/Cisplatin intercalating Gefitinib Treating EGFR Wild NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1.Histological or cytological diagnosis of small-cll lung cancer histology

2.18 years or older

3.Eastern Cooperative Oncology Group (ECOG) Performance Status no more than 2

4.Local stage SCLC without distant metastases

5.After 1st-line chemotherapy (EP or IP) at least 4 cycles

6.After radical radiotherapy for primary tumor and lymph node drainage area:including concurrent or sequence chemoradiotherapy

7.CR or PR assessment by RECIST(1.0) before randomized

8.Haemoglobin 10.0 g/dl, Absolute neutrophil count (ANC) 1.5^9/L, platelets 100 x 10^9/L

9.Total bilirubin 1.5 x upper limit of normal (ULN) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases

10.Creatinine clearance 60ml/min (calculated according to Cockcroft-gault formula)

Exclusion Criteria:

1. Mixed non-small cell lung cancer histology
2. Neck and supraclavicular lymph node metastasis
3. Be allergic to temozolomide or intolerable to radiotherapy
4. Any unstable systemic disease
5. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
disease progression-free survival | 3 years
  the last patient into group for three years or dead

SECONDARY OUTCOMES:
overall survival | 5 years
  the last patients into group for 5 years or dead
side-effects | 3 years
  the last patient into group for 3 years or dead
overall response rate | 3 years
  the last patient into group for 3 years or dead

CONTACTS AND LOCATIONS:
Overall Officials: Jiajia Yu, MD, Study Director — the ethics committee of the first affiliated hospital of Guangzhou MC
Locations (1):
- The first affiliated hospital of Guangzhou MC, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided